CLINICAL TRIAL: NCT06960902
Title: Study of the Determinants of Coronary Atherosclerosis in Familial Hypercholesterolemia
Brief Title: Study of the Determinants of Coronary Atherosclerosis in Familial Hypercholesterolemia (ATHERO-FH Study)
Acronym: ATHERO-FH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: France 2030 program (Unknown); European Union Next Generation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC24_0343; 2025-A00453-46 (Registry Identifier: National number)
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Familial Hypercholesterolemias; Atherosclerotic Cardiovascular Disease (ASCVD)
Keywords: Familial hypercholesterolemia; atherosclerotic cardiovascular disease
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Atherosclerosis

STUDY DESIGN:
Intervention Model Description: Pathophysiology study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): Visit 1: Inclusion Visit: Verification of eligibility criteria. Consent form signing, collection of clinical information, and completion of questionnaires. Fasting blood draw for biological analyses and biobanking. Collection of urine and stool samples (optional). POpmeter (optional), Fibroscan (optional), completion of the CONSTANCES and SF36 questionnaires.
  Visit 2 (30 months): Collection of the CAC score result (dated less than 6 months prior). Collection of clinical information and completion of questionnaires. Fasting blood draw for biological analyses and biobanking. Collection of urine and stool samples (optional). pOpmeter (optional), Fibroscan (optional), completion of the CONSTANCES and SF36 questionnaires.
  Major cardiovascular events will be collected from patients during telephone calls at 1 and 2 years, and during the 30-month visit.
  Interventions: Other: Coronary CT scan with CAC score measurement

INTERVENTIONS:
Other: Coronary CT scan with CAC score measurement — Coronary CT scan with CAC score measurement (on the same day or within 6 months after the inclusion visit).

SUMMARY:
The goal of this study (interventional clinical research not involving a health product) is to assess the prevalence of subclinical coronary atherosclerosis diagnosed by coronary CT angiography in heart failure patients in primary prevention, across different levels of cardiovascular risk defined by coronary artery calcium (CAC) score percentiles (based on data from the MESA study): low risk (≤25th percentile for age, sex, and ethnicity), intermediate risk (25th < CAC ≤ 75th percentile), and high risk (>75th percentile). The Patients will attend an on-site visit at inclusion (and must undergo a coronary CT angiography within 6 months following this visit), will be contacted by phone at 1 year and 2 years, and will return for an on-site visit at 30 months.

ELIGIBILITY:
Inclusion Criteria:

* Person willing to sign the study consent form
* Person affiliated with a current social security scheme
* Person with a definite diagnosis of Familial Hypercholesterolemia, defined by a Dutch Lipid Clinic Network (DLCN) clinical-biological score > 8 and/or an identified causal mutation in the LDL receptor (LDLR) gene, apolipoprotein B100 gene, PCSK9 gene, or apolipoprotein E gene
* Male aged 40 years or older, or female aged 50 years or older
* Ability to understand French for questionnaire completion
* Person not taking any lipid-lowering medication or on a stable dose of lipid-lowering therapy for at least one month prior to inclusion (three months for PCSK9 inhibitors) at Visit 1
* Person not taking any antihypertensive medication or on a stable dose of antihypertensive therapy for at least one month at Visit 1
* Person not taking any antidiabetic medication or on a stable dose of antidiabetic therapy for at least 3 months at Visit 1

Exclusion Criteria:

* Subject with a technical contraindication for coronary CT scan: patient diameter > 70 cm and/or weight > 250 kg
* Patient with a history of atherosclerotic cardiovascular event (myocardial infarction, ischemic heart disease, coronary revascularization, ischemic stroke, carotid endarterectomy, lower limb arterial revascularization)
* Patient allergic to iodinated contrast agents
* Severe renal insufficiency: estimated glomerular filtration rate (eGFR) according to the CKD-EPI formula ≤ 30 ml/min
* Subject with active cancer or in remission for less than 3 years
* Subject who has received oral or intravenous corticosteroid therapy within the last 6 months
* Subject with untreated or poorly controlled hypothyroidism
* Subject receiving immunosuppressive or anticancer therapy
* Subject refusing to participate
* Subject under guardianship, curatorship, or judicial protection, or without social insurance coverage
* Pregnant woman

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2027-03-25 (Estimated); Study Completion 2029-09-25 (Estimated)

PRIMARY OUTCOMES:
Presence of subclinical coronary atherosclerosis | At the time of performing the coronary CT scan
  The criterion defining the presence of subclinical coronary atherosclerosis is the presence of at least one coronary stenosis greater than 50% in a main artery on coronary CT angiography

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - CHU Dijon Bourgogne, Dijon
  - CHRU Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - Hôpital de la Conception, AP-HM, Marseille
  - CHU Nantes, Nantes
  - Hôpital de la Pitié-Salpêtrière, AP-HP, Paris
  - Hôpital Saint-Antoine, AP-HP, Paris
  - CHU Rennes, Rennes
  - CHU Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: Undecided